CLINICAL TRIAL: NCT03801980
Title: Phase 3 Study of SK-1403 ; Double-blinded Parallel Group in Patients With Secondary Hyperparathyroidism Receiving Hemodialysis
Brief Title: Phase 3 Study of SK-1403
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanwa Kagaku Kenkyusho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AJ1004
Record Dates: First submitted 2019-01-08; First posted 2019-01-14 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SK-1403 (Experimental): Patients receive SK-1403 three times a week administered by intravenous bolus injection at the end of each hemodialysis for the whole treatment periods (24 weeks), with individual dose adjustment.
  Interventions: Drug: SK-1403
- Placebo (Placebo Comparator): Patients receive Placebo three times a week administered by intravenous bolus injection at the end of each hemodialysis for the whole treatment periods (24 weeks), with individual dose adjustment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SK-1403 — Patients receive SK-1403 three times a week administered by intravenous bolus injection at the end of each hemodialysis for the whole treatment periods (24 weeks), with individual dose adjustment.
  Arms: SK-1403
Drug: Placebo — Patients receive Placebo three times a week administered by intravenous bolus injection at the end of each hemodialysis for the whole treatment periods (24 weeks), with individual dose adjustment.
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of treatment with SK-1403 for 24 weeks in patients with secondary hyperparathyroidism on maintenance hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Serum PTH>240 pg/mL at the screening
* Serum corrected Ca≧8.4 mg/dL at the screening
* Stable chronic kidney disease patients who undergo hemodialysis or hemodialysis filtration

Exclusion Criteria:

* Primary hyperparathyroidism
* Severe liver disease
* Severe Cardiac disease
* History or family history of long QT syndrome
* Malignant tumor
* Uncontrolled diabetes mellitus
* Uncontrolled hypertension
* History of severe drug allergy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-21 (Actual)

PRIMARY OUTCOMES:
Rate of participants who achieved a mean serum iPTH level of ≥ 60 pg/mL and ≤ 240 pg/mL from 22 to 24 week. | 24 weeks
  Assessed by laboratory test value

SECONDARY OUTCOMES:
Rate of participants who achieved a serum iPTH level of ≥ 60 pg/mL and ≤ 240 pg/mL at each time point. | 24 weeks
  Assessed by laboratory test value
Measured values and Changes from baseline in serum PTH | 24 weeks
  Assessed by laboratory test value; unit of measure (pg/mL)
Measured values and Changes from baseline in Ca | 24 weeks
  Assessed by laboratory test value; unit of measure (mg/dL)
Measured values and Changes from baseline in ionized Ca | 24 weeks
  Assessed by laboratory test value; unit of measure (mEq/dL)
Measured values and Changes from baseline in P | 24 weeks
  Assessed by laboratory test value; unit of measure (mg/dL)
Measured values and Changes from baseline in serum Ca x P product | 24 weeks
  Assessed by laboratory test value

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational site (there may be other sites in this country), Tokyo, Japan

REFERENCES:
- [Derived] Shigematsu T, Koiwa F, Isaka Y, Fukagawa M, Hagita K, Watanabe YS, Honda D, Akizawa T. Efficacy and Safety of Upacicalcet in Hemodialysis Patients with Secondary Hyperparathyroidism: A Randomized Placebo-Controlled Trial. Clin J Am Soc Nephrol. 2023 Oct 1;18(10):1300-1309. doi: 10.2215/CJN.0000000000000253. Epub 2023 Sep 11. PMID 37696667